CLINICAL TRIAL: NCT00956969
Title: Emotional Awareness and Expression Training and Relaxation Training for People With Chronic Headaches
Brief Title: Stress Management for Chronic Headaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Mark A. Lumley, Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WSU0000001
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Headaches
Keywords: headaches; stress management; assertiveness training; relaxation training; emotional expression
MeSH Terms: conditions — Headache | interventions — Gene Expression; Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Anger awareness and expression (Experimental): Training for anger awareness and expression
  Interventions: Behavioral: Anger Awareness and Expression
- Relaxation Training (Active Comparator): Teach patients relaxation training
  Interventions: Behavioral: Relaxation Training
- No-treatment control (No Intervention): Assessment only control condition

INTERVENTIONS:
Behavioral: Anger Awareness and Expression — Teaches patients to recognize, experience, and express emotions
  Arms: Anger awareness and expression
Behavioral: Relaxation Training — Teaches patients relaxation training
  Arms: Relaxation Training

SUMMARY:
This interventional, randomized controlled study seeks to test the effects of a novel emotional awareness and expression intervention against relaxation training or no intervention for college students with chronic headaches. These two interventions are conceptually quite distinct, as the former seeks to activate and process anger, whereas the latter, more commonly used technique, seeks to suppress or avoid it.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate students at Wayne State University who have chronic headaches

Exclusion Criteria:

* Insufficiently frequent headaches
* Uninterested in engaging in a stress management intervention
* Headaches appear due to substance use or head trauma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 147 (Actual)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Headache frequency and severity | baseline, 6-weeks, 6-months

SECONDARY OUTCOMES:
Headache disability | baseline, 6-weeks, 6-months
Mood, self-efficacy, stress symptoms | baseline and 6-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark A. Lumley, Ph.D., Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States